CLINICAL TRIAL: NCT05296525
Title: A Phase I/II Multicenter Study Evaluating the Safety and Efficacy of Allogeneic GDA-201 Natural Killer Cells in Patients With Relapsed/Refractory B Cell Non-Hodgkin Lymphoma
Brief Title: Evaluation of Safety and Efficacy of Allo GDA-201 Natural Killer (NK) Cells in Patients With Relapsed/Refractory B Cell NHL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated by Sponsor.
Sponsor: Gamida Cell ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GC P#01.01.050
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: lymphoma; GDA-201; NK cells; rituximab; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: Dose escalation cohort 1 to reach the maximal tolerated dose, followed by cohort 2 using the recommended Phase II Dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GDA-201 Cohort 1 (Phase I) (Other): Dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Interventions: Drug: GDA-201
- GDA-201 Cohort 2 (Phase II) (Other): RP2D will be administered to all patients.
  Interventions: Drug: GDA-201

INTERVENTIONS:
Drug: GDA-201 — NAM-expanded allogeneic NK cells
  Other Names: Nicotinamide (NAM) NK

SUMMARY:
This is an open-label, non-randomized, interventional, single group assignment study of GDA-201, an allogeneic cryopreserved Natural Killer (NK) cell therapy derived from donor peripheral blood, in combination with rituximab, monoclonal anti-CD20 antibody, for patients with relapsed or refractory B Cell non-Hodgkin lymphoma (NHL).

DETAILED DESCRIPTION:
The study is divided into a phase I dose escalation phase and a phase II expansion phase.

Patients with relapsed or refractory follicular lymphoma (FL) or diffuse large B-cell lymphoma (DLBCL)/high grade B-cell lymphoma (HGBCL) will receive GDA-201 followed by a short course of low-dose interleukin-2 (IL-2). Rituximab will be administered prior to and after GDA-201 infusion.

Phase I: Dose escalation phase The objective of Phase I is to evaluate the safety of GDA-201 in patients with FL, DLBCL/ HGBCL, marginal zone lymphoma or mantle cell lymphoma. The maximal tolerated dose (MTD) and recommended Phase II Dose (RP2D) will be determined based on dose limiting toxicities (DLT).

Phase II expansion phase The objective of the Phase II expansion cohort is to evaluate the safety and efficacy of GDA-201 in two patient cohorts, FL and DLBCL/HGBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have relapsed/refractory FL or HGBCL/DLBCL that has failed conventional therapy defined as follows:

   1. Received at least 2 prior lines of therapy
   2. Transplant ineligible patients allowed assuming they meet criterion a.
   3. Patients who received prior chimeric antigen receptor modified T-cells (CAR-T) cell therapy or are considered ineligible for CAR-T therapy per the investigator's discretion
   4. FL transformed to HGBCL: Must have received at least 1 line of therapy after transformation to DLBCL/HGBCL
2. Patients must be at least 18 years of age
3. Patients must have adequate hematologic, hepatic, renal, cardiac and pulmonary function prior to any study treatment.

Exclusion Criteria:

1. Central Nervous System (CNS) lymphoma
2. Time between previous treatment and first dose of study treatment (rituximab):

   1. Allogeneic hematopoietic stem cell transplantation (HSCT) < 6 months prior to study treatment
   2. Autologous HSCT < 3 months prior to study treatment
   3. CAR-T < 2 months prior to study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Loyola University, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Dana-Farber/Mass General Brigham Cancer Care, Inc., Boston, Massachusetts
  - Henry Ford Medical Center, Detroit, Michigan
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center (MSKCC) - Memorial Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Phase I) -Dose Level 1: Phase I dose escalation with up to 4 dose levels to reach maximum tolerated dose (MTD) and determine recommended Phase II dose (RP2D).
  Dose Level 1: GDA-201 2.5x10^7 cells/kg given in one administration (Day 0)
  Patients followed up to 1y, or death or disease progression, whichever comes first
- Cohort 1 (Phase I) - Dose Level 2: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Dose Level 2: GDA-201 5x10^7 cells/kg given in one (Day 0) or 2 (Day 0 and Day 2) administration(s) Patients followed up to 1y, or death or disease progression, whichever comes first
- Cohort 1 (Phase I) - Dose Level 3: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Dose Level 3: GDA-201 1x10^8 cells/kg given in two administrations (Day 0 and Day 2) Patients followed up to 1y, or death or disease progression, whichever comes first
- Cohort 1 (Phase I) - Dose Level 4: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Dose Level 4: GDA-201 2x10^8 cells/kg given in two administrations (Day 0 and Day 2) Patients followed up to 1y, or death or disease progression, whichever comes first
Period: Dose Level 1 (Week 1 to Week 52)
Arm/Group | Cohort 1 (Phase I) -Dose Level 1 | Cohort 1 (Phase I) - Dose Level 2 | Cohort 1 (Phase I) - Dose Level 3 | Cohort 1 (Phase I) - Dose Level 4
Started | 4 | 0 | 0 | 0
Completed | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Level 2 (Week 23 - Week 75)
Arm/Group | Cohort 1 (Phase I) -Dose Level 1 | Cohort 1 (Phase I) - Dose Level 2 | Cohort 1 (Phase I) - Dose Level 3 | Cohort 1 (Phase I) - Dose Level 4
Started | 0 | 3 | 0 | 0
Completed | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Level 3 (Week 40 - Week 92)
Arm/Group | Cohort 1 (Phase I) -Dose Level 1 | Cohort 1 (Phase I) - Dose Level 2 | Cohort 1 (Phase I) - Dose Level 3 | Cohort 1 (Phase I) - Dose Level 4
Started | 0 | 0 | 3 | 0
Completed | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Level 4 (Week 62 - Week 114)
Arm/Group | Cohort 1 (Phase I) -Dose Level 1 | Cohort 1 (Phase I) - Dose Level 2 | Cohort 1 (Phase I) - Dose Level 3 | Cohort 1 (Phase I) - Dose Level 4
Started | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3
Not completed — Early termination by Sponsor | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- GDA-201 - Cohort 1 (Phase I) - Dose Level 1: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Dose Level 1: GDA-201 2.5x10^7 cells/kg
- GDA-201 - Cohort 1 (Phase I) - Dose Level 2: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Dose Level 2: GDA-201 5x10^7 cells/kg
- GDA-201 - Cohort 1 (Phase I) - Dose Level 3: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Dose Level 3: GDA-201 2.5x10^8 cells/kg
- GDA-201 - Cohort 1 (Phase I) - Dose Level 4: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Dose Level 4: GDA-201 5x10^8 cells/kg
- Total: Total of all reporting groups
Arm/Group | GDA-201 - Cohort 1 (Phase I) - Dose Level 1 | GDA-201 - Cohort 1 (Phase I) - Dose Level 2 | GDA-201 - Cohort 1 (Phase I) - Dose Level 3 | GDA-201 - Cohort 1 (Phase I) - Dose Level 4 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 1 | 6
  >=65 years | 2 | 1 | 2 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 6
  Male | 2 | 2 | 1 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 3 | 3 | 3 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 3 | 13
Patient diagnosis [Count of Participants; unit: Participants]
  Follicular lymphoma | 1 | 0 | 0 | 1 | 2
  Diffuse large B-cell lymphoma | 2 | 1 | 0 | 2 | 5
  High grade B-cell lymphoma | 1 | 1 | 1 | 0 | 3
  Marginal zone lymphoma | 0 | 1 | 1 | 0 | 2
  Mantle cell lymphoma | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Safety as Determined by Dose Limiting Toxicities (DLTs)
Description: DLTs defined as one of the following within the first 28 days of the first dose of GDA-201 by the NCI-CTCAE v 5.0. acute graft-versus-host disease (aGvHD) will be assessed according to the Consensus Conference on aGvHD grading:
  Steroid refractory Grade II aGvHD, defined as GvHD that does not respond to at least 1 mg/kg/day or equivalent of prednisone within 7 days of initiating therapy Grade III or IV aGvHD Grade 4 infusion reaction Grade 4 or 5 related adverse event (AE) Grade 3 or above cardiac, central nervous system or pulmonary adverse event. Any Grade 3 or above non-hematologic adverse event that does not resolve to Grade 2 or below within 72 hours, except for renal or hepatic adverse events which may take up to 7 days to resolve Treatment emergent ≥Grade 3 autoimmune disorder Grade 3 or above allergic reaction that does not recover to Grade II or below within 24 hours Grade 4 cytopenia lasting beyond Day 42 (the 28-day DLT observation period will be extend
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Groups:
- GDA-201 - Cohort 1 (Phase I) - Dose Level 3: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Dose Level 3: GDA-201 1x10^8 cells/kg
- GDA-201 - Cohort 1 (Phase I) - Dose Level 4: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended Phase II dose (RP2D).
  Dose Level 2: GDA-201 5x10^8 cells/kg
Arm/Group | GDA-201 - Cohort 1 (Phase I) - Dose Level 1 | GDA-201 - Cohort 1 (Phase I) - Dose Level 2 | GDA-201 - Cohort 1 (Phase I) - Dose Level 3 | GDA-201 - Cohort 1 (Phase I) - Dose Level 4
Number analyzed (Participants) | 4 | 3 | 3 | 3
Participants
  Patients who experienced dose limiting toxicities (DLTs) | 0 | 0 | 0 | 0
  Patients who did not experience DLT | 3 | 3 | 3 | 2
  Patients not evaluable for DLT | 1 | 0 | 0 | 1

2. Primary Outcome: Phase II: Overall Response Rate
Description: Patients will be assessed after the infusion of GDA-201 for level of response.
Time Frame: up to 1 year
Population: Study was early terminated by Sponsor prior to initiation of the phase II
Groups:
- GDA-201 Cohort 2 (Phase II): RP2D will be administered to all patients.
  GDA-201: Nicotinamide(NAM)-expanded allogeneic NK cells
Arm/Group | GDA-201 Cohort 2 (Phase II)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected between initiation of study treatment until end of study participation for each patient (up to one year, or death/disease progression/early termination, whichever came first).
Description: Any event after written informed consent has been obtained and prior to study treatment initiation was recorded as medical history unless the event was directly related to a screening procedure, in such case it was considered an Adverse Event (AE)/Serious adverse event (SAE)
Groups:
- GDA-201 Cohort 1 (Phase I) - Dose Level 1: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended phase II dose (RP2D).
  Dose Level 1: GDA-201 2.5x10^7 cells/kg given in one administration (Day 0)
- GDA-201 Cohort 1 (Phase I) - Dose Level 2: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended phase II dose (RP2D).
  Dose Level 2: GDA-201 5x10^7 cells/kg given in one (Day 0) or two (Day 0 and +2) administrations
- GDA-201 Cohort 1 (Phase I) - Dose Level 3: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended phase II dose (RP2D).
  Dose Level 3: GDA-201 5x10^7 cells/kg given in two administrations (Day 0 and +2)
- GDA-201 Cohort 1 (Phase I) - Dose Level 4: Phase I dose escalation with up to 4 dose levels to reach MTD and determine recommended phase II dose (RP2D).
  Dose Level 4: GDA-201 5x10^7 cells/kg given in two administrations (Day 0 and +2)
Arm/Group | GDA-201 Cohort 1 (Phase I) - Dose Level 1 | GDA-201 Cohort 1 (Phase I) - Dose Level 2 | GDA-201 Cohort 1 (Phase I) - Dose Level 3 | GDA-201 Cohort 1 (Phase I) - Dose Level 4
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDA-201 Cohort 1 (Phase I) - Dose Level 1 (N=4) | GDA-201 Cohort 1 (Phase I) - Dose Level 2 (N=3) | GDA-201 Cohort 1 (Phase I) - Dose Level 3 (N=3) | GDA-201 Cohort 1 (Phase I) - Dose Level 4 (N=3)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDA-201 Cohort 1 (Phase I) - Dose Level 1 (N=4) | GDA-201 Cohort 1 (Phase I) - Dose Level 2 (N=3) | GDA-201 Cohort 1 (Phase I) - Dose Level 3 (N=3) | GDA-201 Cohort 1 (Phase I) - Dose Level 4 (N=3)
Abdominal distention (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (7) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (2) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Culture urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Hepatobiliary procedural complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (4) | 1 (2) | 2 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (11) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (9) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (6) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Pain (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 2 (4) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (3) | 0 (0) | 1 (3) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT05296525/Prot_SAP_001.pdf